CLINICAL TRIAL: NCT06026280
Title: Developing an App-based Behavioral Intervention to Help Depressed Individuals Return to Work
Brief Title: Depression Return to Work Intervention
Acronym: DRIVEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inspiration at Work (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R42MH127971 (NIH)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Job Stress; Distress, Emotional
Keywords: depression; unemployment
MeSH Terms: conditions — Occupational Stress; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Job-Search Program (Placebo Comparator): 6 weeks of self-guided job-seeking
  Interventions: Other: Career Resources
- DRIVEN App-Based Program (Experimental): 6 weeks of job-seeking guided by the DRIVEN curriculum
  Interventions: Behavioral: DRIVEN Application

INTERVENTIONS:
Behavioral: DRIVEN Application — Participants will complete the six-week DRIVEN program, which includes a smartphone application and job coaching.
  Arms: DRIVEN App-Based Program
Other: Career Resources — Participants will receive weekly information about job-searching skills and resources from a study coordinator for six weeks.
  Arms: Conventional Job-Search Program

SUMMARY:
This study is a randomized controlled trial to test the effectiveness of a mobile app-based program aimed to help individuals with unemployment-related emotional distress return to work.

DETAILED DESCRIPTION:
This study will compare two different approaches to reducing unemployment-related emotional distress. Participants will be involved in the study for a total of 22 weeks. During the first 6 weeks, participants will complete activities relating to either the mobile-app based program or the self-guided job-seeking program. The study team will follow up with participants at 8 weeks after the program is completed and at 16 weeks after the program is completed. Participants will also be asked to complete questionnaires before starting the program, during the program, after they complete the program, and at the follow-up visits. The questionnaires will be about the participant's mood, job seeking behavior, and related emotional experiences.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Currently unemployed and actively searching for work
* Prior to unemployment, were employed full-time (35 hours per week or more) for at least 1 year
* Prior to unemployment, received an individual highest salary of $100,000 or less
* Owns an iPhone or Android Phone
* Willing and able to provide informed consent
* Has a minimum depression score according to the PROMIS depression scale
* Able to communicate in English (verbal and written)

Exclusion Criteria:

* Current moderate or severe alcohol/substance use disorders
* Current symptoms of mania or psychosis
* Currently employed, retired, or a full or part-time student

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Job Search Behavior (JSB) Scale | Baseline; Each week of the program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  10-item scale to assess the frequency that a person performs certain job seeking behaviors within a week. Each item has 5 answer options (from 0 times to 6 or more times). A higher score indicates that someone performs more job seeking behaviors each week.

SECONDARY OUTCOMES:
Job Search Self Efficacy (JSSE) Scale | Baseline; Week 3 of program; Week 6 of program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  20-item scale to assess someone's confidence in performing job seeking behaviors and achieving job seeking outcomes. Each item has 5 answer options (from 1 to 5). Raw scores of items from each domain are averaged to produce a final domain score between 1 and 5. A higher score indicates that someone is more confident in performing a job seeking behavior or achieving a job seeking outcome, depending on the domain.
The Inventory of Depression and Anxiety Symptoms (IDAS) - Social Anxiety Subscale | Baseline; Week 3 of program; Week 6 of program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  6-item scale to assess social anxiety symptoms. Each item has 5 answer options (from 1 to 5). A higher score indicates a greater presence of that symptom within the past two weeks.
Patient Reported Outcome Measures Information System (PROMIS) Depression Scale | Baseline; Each week of the program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  8-item scale to assess depression. Each item has 5 answer options (from 1 to 5). Minimum score = 8; maximum score = 40. A higher score indicates a greater presence of depressive symptoms.
Patient Reported Outcome Measures Information System (PROMIS) Positive Affect Scale | Baseline; Each week of the program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  15-item scale to assess positive affect. Each item has 5 answer options (from 1 to 5). Minimum score = 15; maximum score = 75. A higher score indicates a greater presence of positive affect.
Patient Reported Outcome Measures Information System (PROMIS) Meaning and Purpose Scale | Baseline; Week 6 of program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  8-item scale to assess meaning and purpose in someone's life. Each item has 5 answer options (from 1 to 5). Minimum score = 8; maximum score = 40. A higher score indicates a greater sense of meaning and purpose.
Cognitive Behavioral Avoidance Scale (CBAS) | Baseline; Week 5 of program; Week 6 of program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  31-item scale to assess what strategies someone uses to deal with situations and problems, with strategies falling into the domains of behavioral-social, cognitive-nonsocial, cognitive-social, and behavioral-nonsocial. Each item has 5 answer options (from 1 to 5). Raw scores of items from each domain are summed to produce a final domain score. A higher score indicates a greater presence of that coping strategy in someone's life.
Behavioral Activation for Depression Scale (BADS) | Baseline; Week 5 of program; Week 6 of program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  9-item scale to assess behavioral activation. Each item has 7 answer options (from 0 to 6). Minimum score = 0; maximum score = 54. A higher score indicates higher activation.
Cognitive Flexibility Inventory (CFI) | Baseline; Week 5 of program; Week 6 of program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  20-item scale to assess cognitive flexibility. Each item has 7 answer options (from 1 to 7). Minimum score = 20; maximum score = 140. A higher score indicates more cognitive flexibility.
Participant Global Impression of Change (PGIC) | Week 6 of program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  To assess participant's impression of change in their depression since the start of the intervention. This scale is 1-item. Minimum score = 1; maximum score = 5. A higher score indicates the best change since starting the intervention.
System Usability Scale (SUS) | Week 1 of program; Week 6 of program
  10-item measure to assess the usability of the program. Each item has 5 answer options (from 1 to 5). Minimum raw score = 0; maximum raw score = 40. Raw scores are multiplied by 2.5 to give a final score of 0 (representing the worst usability) to 100 (representing the best usability).
Job Status Questionnaire | Each week of the program; Follow-up (8 weeks after program); Follow-up (16 weeks after program)
  Measure to assess whether or not someone obtained a job throughout the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra R. Levit, Principal Investigator — Inspiration at Work; Stewart A. Shankman, PhD, Principal Investigator — Northwestern University, Department of Psychiatry and Behavioral Sciences; James W. Griffith, PhD, Principal Investigator — University of Chicago
Locations (1):
- Inspiration at Work, Inc., Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danielson EC, Saturday M, Leonard S, Levit A, Graham AK, Marquez M, Alperin K, Shankman SA, Griffith JW. Efficacy of a Mobile App-Based Behavioral Intervention (DRIVEN) to Help Individuals With Unemployment-Related Emotional Distress Return to Work: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Nov 26;13:e62715. doi: 10.2196/62715. PMID 39589786

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT06026280/SAP_000.pdf